CLINICAL TRIAL: NCT07332923
Title: Development of a Machine Learning-Based Nomogram for Predicting HIF-2α Expression Levels in Clear Cell Renal Cell Carcinoma
Brief Title: Predicting HIF-2α Levels in Clear Cell Kidney Cancer Using Machine Learning
Status: Active, not recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: MRCTA,ECFAH OfFMUI2024]639
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Renal Clear Cell Carcinoma; HIF-2α; Radiomics; Nomogram
Keywords: Nomogram; Radiomics; HIF-2α; Renal clear cell carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project aims to conduct a multicenter retrospective study to collect clinical, CT imaging, and pathological data from patients. A comprehensive data management system will be established, and radiomic features will be extracted to integrate and analyze multicenter data. We will develop a predictive model based on CT radiomic features and perform both internal and external cohort validation. The model will predict HIF-2α expression levels and clinically relevant prognostic factors in ccRCC, enabling precise identification of patient populations responsive to the HIF-2α antagonist Belzutifan, thereby facilitating personalized treatment decisions, minimizing unnecessary therapeutic risks, and ultimately improving patient quality of life and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed clear cell renal cell carcinoma (ccRCC)
* Availability of comprehensive clinical, pathological, and follow-up information
* Access to preoperative non-contrast and contrast-enhanced CT images through the PACS database
* Adequately preserved pathological slides for subsequent immunohistochemical (IHC) or tissue microarray analysis
* Minimum of one post-treatment follow-up with documented treatment response or efficacy evaluation

Exclusion Criteria:

* Patients considered ineligible for treatment owing to severe comorbid conditions or inability to undergo any therapeutic intervention
* Patients with concurrent malignancies, including prior treatment for other cancers or presence of untreated active malignancies
* Patients with inadequate CT image quality or missing imaging data
* Patients with missing or incomplete clinical, pathological, or follow-up information

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with histologically confirmed renal cell carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
HIF-2α Expression Levels in Clear Cell Renal Cell Carcinoma | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- first hospital affiliated of Fujian medical university, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided